CLINICAL TRIAL: NCT03203239
Title: Vasodilatory Effects of Light on Peripheral Artery Disease
Brief Title: Red Light Treatment in Peripheral Artery Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Nicole Lohr, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 29388
Record Dates: First submitted 2017-06-27; First posted 2017-06-29 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Artery Disease; Claudication, Intermittent; Vasodilation
Keywords: red light; vasodilation; nitric oxide
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Aneurysm | interventions — perflutren

STUDY DESIGN:
Intervention Model Description: This is a single group study in which the subject undergoes a single exposure to red light.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Red Light treatment (Experimental): This is a single arm design. All subjects will be enrolled to have peripheral blood flow measured before, during, and after red light exposure.
  Interventions: Device: Red Light (670 nm energy); Drug: Octafluoropropane

INTERVENTIONS:
Device: Red Light (670 nm energy) — Light Emitting Diode light source (670 nm wavelength with output up to 75mW/cm2) will be placed over the gastrocnemius muscle. The light will be on for 5 minutes.
Drug: Octafluoropropane — All subjects will undergo infusion of octafluoropropane to measure peripheral blood flow.
  Other Names: Definity

SUMMARY:
Subjects with a known diagnosis of peripheral artery disease as measured by an abnormal ankle brachial index (<.9 or >1.1) will undergo a single 5 min exposure of 670 nm light, 1 cm above the gastrocnemius muscle. Blood flow will be measured by infusion of ultrasound contrast and subsequent acquisition of ultrasound images. 2 blood samples will be collected for measurement of nitric oxide metabolites.

DETAILED DESCRIPTION:
The intent of this protocol is to measure blood flow in the gastrocnemius muscle in patients with documented peripheral artery disease before and after exposure to 670 nm light energy. The study consists of one visit. Blood flow measurement will be performed using contrast enhanced ultrasound, a method by which ultrasound contrast is continuously infused into the blood stream. Ultrasound records images in the area of interest and flow is related to the intensity of the contrast in each image. Blood will be drawn to measure nitric oxide metabolites. The study is designed to consist of one visit. However, if the protocol changes or the data quality initially collected is uninterpretable, subjects may be asked to return to allow for a standard methodology across all participants. In this case, the subjects who are asked to return will be subject to the same informed consent process a second time. The two visits will be at least one week apart to further reduce the already minimal risks of the study. This will also limit the number of study participants required to gather the necessary data to complete the study, thereby limiting the risks of the study to a smaller number of participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be subjects between the ages of 18 and 85 who have been diagnosed with peripheral artery disease. Men and women will be recruited for participation. All ethnicities will be included in this study.

Diagnosis of peripheral artery disease is defined as an Ankle Brachial index of <0.9 or greater than 1.1 either at rest or during treadmill exercise.

Exclusion Criteria:

* Exclusionary criteria include age under 18 years and over 85 years, those who are unable to understand the consent process , those who cannot read or speak English, active pregnancy, hypersensitivity to perflutren contrast agents, pulmonary hypertension, active illicit drug use, untreated blood pressure over 160/95, sickle cell disease, or a history of intracardiac shunt. Additional exclusion criteria neurological diseases such as spinal stenosis, unspecified pain disorders, and any uncontrolled medical conditions.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in blood flow | Baseline, 5 min of light, and up to 1 min after discontinuation of light
  Video intensity units from contrast images will be converted to ml/min/g tissue

SECONDARY OUTCOMES:
Changes in nitric oxide metabolites | Baseline and 1 min after discontinuation of light
  NO measurement by ozone chemiluminescence

CONTACTS AND LOCATIONS:
Overall Officials: Nicole L Lohr, MD,PHD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No